CLINICAL TRIAL: NCT02135874
Title: A Phase 2 Study of Clofarabine, Idarubicin, Cytarabine, Vincristine, and Corticosteroids for Patients With Newly Diagnosed or Relapsed Mixed Phenotype Acute Leukemia
Brief Title: Clofarabine, Idarubicin, Cytarabine, Vincristine Sulfate, and Dexamethasone in Treating Patients With Newly Diagnosed or Relapsed Mixed Phenotype Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0073; NCI-2014-02322 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0073 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Acute Bilineal Leukemia; Acute Biphenotypic Leukemia; Acute Leukemia of Ambiguous Lineage; Acute Undifferentiated Leukemia; Mixed Phenotype Acute Leukemia; Mixed Phenotype Acute Leukemia, B/Myeloid, Not Otherwise Specified; Mixed Phenotype Acute Leukemia, T/Myeloid, Not Otherwise Specified; Recurrent Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute | interventions — Clofarabine; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Idarubicin; Rituximab; CT-P10; Sorafenib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): See Detailed Description.
  Interventions: Drug: Clofarabine; Drug: Cytarabine; Drug: Dexamethasone; Drug: Idarubicin; Biological: Rituximab; Drug: Sorafenib; Drug: Sorafenib Tosylate; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Clofarabine — Given IV
  Other Names: Clofarex; Clolar
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43-9006; Bay-439006
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well clofarabine, idarubicin, cytarabine, vincristine sulfate, and dexamethasone work in treating patients with mixed phenotype acute leukemia that is newly diagnosed or has returned after a period of improvement (relapsed). Drugs used in chemotherapy, such as clofarabine, idarubicin, cytarabine, vincristine sulfate, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the response rate of the chemotherapy regimen in patients with mixed phenotype acute leukemia.

SECONDARY OBJECTIVE:

I. To evaluate the durability of response, the overall and event-free survival rates, and the safety profile of the regimen.

OUTLINE:

INDUCTION THERAPY: Patients receive clofarabine intravenously (IV) over 60 minutes on days 1-4 or 1-3; idarubicin IV over 30-60 minutes on days 1-3 or 1-2; cytarabine IV over 2 hours on days 1-4; vincristine sulfate IV over 15-30 minutes on days 1, 8, and 15; and dexamethasone IV over 10-30 minutes on days 1-4 and 15-18. Patients with a certain type of leukemia may receive rituximab IV over 4-6 hours on days 1 and 8 or sorafenib tosylate orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients receive clofarabine IV over 60 minutes on days 1-3 or 1-2; idarubicin IV over 30-60 minutes on days 1-2; cytarabine IV over 2 hours on days 1-3 or 1-2; vincristine sulfate IV over 15-30 minutes on days 1, 8, and 15; and dexamethasone IV over 10-30 minutes on days 1-4 and 15-18. Patients with a certain type of leukemia may receive rituximab IV over 4-6 hours on days 1 and 8 of cycles 1-3 or sorafenib tosylate PO BID on days 1-28 of cycle 1-6 and beyond. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent document
* Newly diagnosed or relapsed mixed phenotype acute leukemia (MPAL), which for this protocol, will be defined as follows: bone marrow result interpreted by the reading pathologist (or tissue biopsy for cases of extramedullary disease) as: biphenotypic leukemia, bilineal leukemia, undifferentiated leukemia, mixed lineage leukemia, leukemia of ambiguous lineage, T/myeloid leukemia, B/myeloid leukemia, or other diagnosis indicating the presence of multiple lineages within the cell population
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3 at study entry
* Adequate organ function as outlined below (unless due to leukemia)
* Serum creatinine =< 3 mg/dL
* Total bilirubin =< 2.5 mg/dL
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and/or aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper limit of normal (ULN) or =< 5 x ULN if related to disease
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days; women of childbearing potential and men must agree to use contraception at study entry and for the duration of active study treatment
* Cardiac ejection fraction >= 40% (by either cardiac echocardiogram [echo] or multi gated acquisition [MUGA] scan); documentation of recent (=< 6 months from screening) outside reports is acceptable
* If newly diagnosed, prior therapy with hydrea and/or steroid and the use of a single or a two day dose of cytarabine (up to 3 g/m^2), for emergency use up to 24 hours prior to start of study therapy is allowed

Exclusion Criteria:

* Breast feeding females
* Patients with active, uncontrolled infections
* Patients with active secondary malignancy will not be eligible unless approved by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 59 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 7
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Participants Complete Response
Description: Response is Complete Response (CR) is Neutrophil count >/= 1.0 x 10^9/L, . Platelet count >/= 100 x 10^9/L, Bone marrow aspirate < 5% blasts, No extramedullary leukemia.
Time Frame: Up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 16
Participants | 9

2. Secondary Outcome: 4-week Mortality Rate
Description: Number of participants who died after 4 weeks of treatment.
Time Frame: At 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 8 years
Arm/Group | Treatment (Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 3/16
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy) (N=16)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Central Line blood stream Infection (Infections and infestations) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5)
Right Atrial Thrombus removal (Surgical and medical procedures) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Thromboembolic Event (Vascular disorders) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Sepsis Tracheal Aspiration (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy) (N=16)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fluid Imbalance (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transaminitis (Metabolism and nutrition disorders) | 5 (5)
Pain Ear (Ear and labyrinth disorders) | 1 (1)
Pain Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (General disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Elevated INR (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Bruise (General disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Immunosuppression (Immune system disorders) | 2 (2)
Cellulitis- L great toe (Infections and infestations) | 1 (1)
Facial swelling (General disorders) | 2 (2)
Infection skin lesion (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Elevated Creatinine (Blood and lymphatic system disorders) | 1 (1)
Paralytic Ileus (Gastrointestinal disorders) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT02135874/Prot_SAP_000.pdf